CLINICAL TRIAL: NCT05386927
Title: Clinical Study of a New Technology System for Early Diagnosis and Screening of GDM Based on Multiomics
Brief Title: Early Diagnosis of GDM by Multiomics
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Women's Hospital School Of Medicine Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: IRB-20210293-R
Record Dates: First submitted 2022-05-15; First posted 2022-05-23 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-07

CONDITIONS: Gestational Diabetes Mellitus
MeSH Terms: conditions — Diabetes, Gestational | interventions — Specimen Handling

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, urine and saliva from pregnant women will be collected for testing
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- GDM group: Pregnant women with positive OGTT results at 24-28 gestational weeks
  Interventions: Other: Questionnaire survey and specimen collection
- Control group: Pregnant women with negative OGTT results at 24-28 gestational weeks, and had baseline data that matched those in the GDM group
  Interventions: Other: Questionnaire survey and specimen collection

INTERVENTIONS:
Other: Questionnaire survey and specimen collection — A questionnaire survey was conducted when pregnant women were enrolled in the first trimester, and blood, urine, saliva and other specimens were collected.

SUMMARY:
Gestational diabetes mellitus (GDM) is prone to cause a variety of adverse pregnancy outcomes, and has potential harm to the short-term and long-term health of both mothers and infants. However, its diagnosis mainly relies on oral glucose tolerance test (OGTT) at 24-28 weeks of gestation, so it is often diagnosed in the second and third trimester, and may be too late to intervene. Therefore, advancing the diagnostic window period of GDM is the key to the prevention and treatment of GDM and its complications. It is urgent to establish a new technology for the early diagnosis and screening of GDM with high detection rate and accuracy. Based on literature survey and previous studies, this study found that the combined analysis of metabolomics and lipidomics may have broad clinical application prospects in the early diagnosis and screening of GDM. It is hoped that a set of new techniques based on multi-omics for early diagnosis and screening of GDM can be constructed, providing a feasible and effective tool for early detection and treatment of GDM in clinical.

ELIGIBILITY:
Inclusion Criteria:

* Plan to have routine prenatal examinations and give birth in the research center
* First trimester
* Singleton pregnancy
* Without pregnancy complications
* Willing to cooperate with the hospital to follow up

Exclusion Criteria:

* Have diseases that affect metabolic function or even threaten the life of the mother and fetus before pregnancy, such as diabetes, heart disease, liver and kidney diseases, thyroid diseases with drug, autoimmune diseases, malignant tumors, AIDS, etc.
* Fetus has a known deformity or genetic defects
* Incomplete clinical data

Ages: 20 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: This project intends to recruit pregnant women who go to the research center for routine prenatal examination and OGTT screening.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Salivary metabolomics | First trimester (9-14 gestational weeks)
  The differential salivary metabolism molecules in saliva were detected by the self-developed detection chip, and the markers related to GDM in early pregnancy were screened. Specimens were collected during the first trimester.
Serum lipidomics | First trimester (9-14 gestational weeks)
  The differential serum lipid molecules in serum were detected by the self-developed detection chip, and the markers related to GDM in early pregnancy were screened. Specimens were collected during the first trimester.
Urine metabolomics | First trimester (9-14 gestational weeks)
  The differential urine metabolism molecules in urine were detected by the self-developed detection chip, and the markers related to GDM in early pregnancy were screened. Specimens were collected during the first trimester.

CONTACTS AND LOCATIONS:
Overall Officials: Zhaoxia Liang, Prof., Study Director — Women's Hospital School Of Medicine Zhejiang University
Locations (1):
- Women's Hospital School Of Medicine Zhejiang University, Hangzhou, Zhejiang, China